CLINICAL TRIAL: NCT01082666
Title: Phase 4 Study of Continuous Control of Tracheal Cuff Pressure and Microaspiration in Critically Ill Patients
Brief Title: Continuous Control of Tracheal Cuff Pressure and Microaspiration in Critically Ill Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008_53/0919; 2009-A00431-56 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2010-02-05; First posted 2010-03-08 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Critically Ill
Keywords: Cuff pressure; microaspiration; pepsin; VAP; Mechanical ventilation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous control (Experimental): Continuous control of cuff pressure using a pneumatic device
  Interventions: Device: Continuous control of cuff pressure
- Manual control (Active Comparator): Manual control of cuff pressure is a routine practice in ICU patients
  Interventions: Device: Manual control of cuff pressure

INTERVENTIONS:
Device: Continuous control of cuff pressure — Continuous control of cuff pressure using a pneumatic device (Nosten, Leved, France)
  Other Names: Automatic control of cuff pressure (Rusch, Kernen, Germany)
  Arms: Continuous control
Device: Manual control of cuff pressure — Manual control of cuff pressure is a routine practice in ICU patients
  Other Names: Manual manometer
  Arms: Manual control

SUMMARY:
We hypothesized that continuous control of tracheal cuff pressure would reduce microaspiration of gastric content as determined by pepsin level in tracheal aspirate.

DETAILED DESCRIPTION:
Randomized controlled open label study, performed in a 10-bed ICU. All patients intubated with a PVC-cuffed tracheal tube and receiving enteral nutrition who require at least 48 h of mechanical ventilation are eligible. Patients receive continuous control of cuff pressure using a pneumatic device (intervention group) or manual control using a manometer (control group). Target cuff pressure is 25 cmH2O.

In all patients, pepsin is measured in tracheal aspirate during a 48-h period after inclusion, as proxy for gastric content aspiration. In addition tracheobronchial colonization and ventilator associated pneumonia rates will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* age > or = 18 years
* tracheal intubation using a polyvinylchloride tube
* predictible duration of mechanical ventilation > 48 h
* enteral nutrition

Exclusion Criteria:

* refuse to participate to the study
* no informed consent
* contra-indication for semirecumbment position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pepsin level in tracheal aspirate | 48 h after randomization

SECONDARY OUTCOMES:
Ventilator-associated pneumonia, tracheobronchial colonization, tracheal ischemic lesions | day 28 after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Alain Durocher, MD, Study Director — CHRU de Lille; Malika Balduyck, MD, Study Director — CHU de Lille; Farid Zerimech, MD, Study Director — CHU de Lille
Locations (1):
- ICU, Calmette Hospital, University Hospital of Lille, Lille, Nord, France